CLINICAL TRIAL: NCT06615505
Title: ASCEND: A Randomized, Double Blind, Sham-Controlled, Multi-Center Phase I/II Clinical Trial to Evaluate the Safety and Effectiveness of VIA Disc NP, a Supplement for Degenerated Intervertebral Discs
Brief Title: ASCEND: A Clinical Trial to Evaluate the Safety and Effectiveness of VIA Disc NP, a Supplement for Degenerated Intervertebral Discs
Acronym: ASCEND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VIVEX Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: VIA-2024-001
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Degenerative Disc Disease; Disc Degeneration; Lumbar Discogenic Pain
Keywords: Degenerative Disc Disease; Lumbar Discogenic Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: At the 12-week follow-up, all participants will remain blinded and will be given the option to be considered for crossover. Only participants allocated to the needle sham control group will be given the option to crossover into the VIA Disc NP group at the 12-week visit if they meet the following requirement:
  The participant has not experienced at least a 30% reduction in pain severity as determined by their 12-week VAS score
  Sham participants who crossover into the VIA Disc NP group will receive an injection of VIA Disc NP and continue in the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The following individuals should be blinded in the ASCEND Clinical Trial:
  Participants: when randomized into the trial, the patient will consent to be blinded to the type of treatment they will receive
  Outcome assessors:
  * Clinicians (sub-Is) completing the physical or neurological examination
  * Study coordinator administering patient-reported outcomes and collecting other participant data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIA Disc NP (Active Comparator)
  Interventions: Other: VIA Disc NP
- Sham Arm (Sham Comparator)
  Interventions: Other: Sham Injection

INTERVENTIONS:
Other: VIA Disc NP — Participants will receive a single dose, intradiscal injection of 100 mg of VIA Disc NP mixed with sterile saline according to product Instructions for Use (IFU) and administered to the affected level(s), L1-S1 (1 or 2 levels).
  Arms: VIA Disc NP
Other: Sham Injection — Participants will receive the sham procedure at 1 or 2 levels.
  The procedure will be identical to the investigational procedure with the following exception: A 20G spinal needle will be carefully inserted through the skin and muscle of the back but WILL NOT penetrate the annulus fibrosus of the intervertebral disc.
  Arms: Sham Arm

SUMMARY:
VIA Disc NP is an off-the-shelf minimally processed human nucleus pulposus tissue allograft intended to supplement degenerated intervertebral discs.

The study is a randomized, double-blind, sham-controlled, multi-center study in participants with symptomatic lumbar intervertebral disc degeneration (> 6 months) and unresponsive to conservative therapy for at least 3 months. Participants will be randomized on a 1:1 basis to receive either a single VIA Disc NP intradiscal injection at 1 or 2 levels or a sham procedure at 1 or 2 levels.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 22 to 85 years old
2. Diagnosis of early to moderate DDD, Modified Pfirrmann Grade 3-7
3. Chronic axial midline low-back pain with or without referred non-radicular leg pain for at least 6 months prior to screening; unresponsive to at least 3 months of conservative care
4. Positive hip flexion test as confirmed with the Neurologic Exam indicating positive provocation with sustained hip flexion at the time of screening
5. Demonstrated intolerance to sitting for more than 30 minutes at a time based on self-report or assessed by a qualified healthcare professional at the screening visit
6. Low-back pain severity score of ≥ 40 to ≤ 90 mm on the VAS at the time of Screening
7. ODI score of ≥ 40 to ≤ 80 at the time of Screening

Key Exclusion Criteria:

1. Contraindication to MRI for any reason
2. Contraindications to the proposed sedation/anesthetic protocol
3. Symptomatic involvement of more than two lumbar discs
4. Fracture of the spine, previous lumbar spine surgery or previous treatment of the target disc(s)
5. Grade 2 or higher spondylolisthesis at the target disc, lumbar spondylitis or other undifferentiated spondyloarthropathy, or Type III Modic changes around the target disc
6. Clinical suspicion of a full thickness annular tear at the target disc or other abnormal disc morphology
7. Clinical suspicion of facet pain as primary pain generator
8. Women who are pregnant or breastfeeding at the time of enrollment and/or plan to become pregnant during the study. Pregnancy is confirmed by:

   * A positive pregnancy test during the screening visit
   * Self-reported pregnancy
9. Women of childbearing potential (WOCBP) who are not using a reliable form of contraception (as determined by the Investigator)

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint - Proportion of participants achieving MCID in VAS score from Baseline to 26 weeks. | Baseline to 26 Weeks
  A comparison of the proportion of participants who show a minimally clinically important difference (MCID), defined as at least a 30% reduction in back pain VAS score from baseline to 26 weeks (6 months), in the VIA Disc NP group to that in the sham-control group.
Primary Safety Endpoint - Proportion of participants reporting Treatment-related AEs at 12 weeks | Baseline to 12 weeks
  The proportion of participants that experience one or more treatment-related (including procedure) adverse events in the VIA Disc NP group compared to the sham-control group at 12 weeks (3 months) as determined by the Principal Investigator.

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Genesis Research Services Pty Ltd, Broadmeadow, New South Wales
  - Australian Medical Research, Hurstville, New South Wales
  - Sydney Pain Research Centre, Wahroonga, New South Wales
  - Cercare Clinical Research, Wayville, South Australia
  - Monash Clinical Research Pty Ltd, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No